CLINICAL TRIAL: NCT03942471
Title: The Effects of Learning Mindfulness Based Stress Reduction on Psychosocial Variables and HbA1c in Adolescents With Type 1 Diabetes
Brief Title: Mindfulness for Adolescents With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duquesne University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2015/10/14
Record Dates: First submitted 2019-03-29; First posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: between and within group repeated measures design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Mindfulness Based Stress Reduction (Other): Six Modules each delivering an important principle of Mindfulness Based Stress Reduction
  Interventions: Behavioral: Mindfulness Based Stress Reduction
- Control Group (No Intervention): Wait Group - received no mindfulness teaching

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction — Mindfulness-Based Stress Reduction (MBSR) is a well-defined and systematic patient-centered educational approach which provides training in mindfulness meditation to teach adolescents with Type 1 diabetes to take better care of themselves and live healthier and more adaptive lives by learning to become more connected to the present moment through the use of breath and training for awareness of the moment.
  Other Names: MBSR
  Arms: Intervention Mindfulness Based Stress Reduction

SUMMARY:
Adolescents with Type 1 Diabetes will be invited to the Mindfulness study. They will be randomly assigned to a Control or Active Group. The Active Group will learn Mindfulness Based Stress Reduction (MBSR) through an online website designed to teach the basic principles of MBSR in six week-long modules. They will be measured in three main areas: before learning the intervention, directly after learning it and 3 months after learning it to determine any changes in their Mindful attention awareness, Diabetes Quality of Life and HbA1c. The Control Group will also take the questionnaires at the beginning of the study, 6 weeks after it begins and then 3 months from the beginning to obtain data for all three time points when they have not received access to the modules/intervention.

DETAILED DESCRIPTION:
Research Design and Procedures This study will utilize a between group repeated measures design to measure the effects of the learned MBSR intervention over time. MBSR will be the independent variable. Dependent variables include mindfulness, diabetic quality of life and HbA1c. Adolescents with Type 1 diabetes will be randomly assigned to an intervention group or a wait list/control group that will be taught MBSR after all data has been collected. The study will utilize a 2 (experimental versus wait-list control group) by 3 (pretest [Time 1], posttest [Time 2], and 3 month follow-up [Time 3]) to examine within and between group differences overtime on two psychosocial measures including mindfulness and quality of life. The physiological measure understudy, HbA1c, reflects glucose control over the previous three month period and will be measured at Time 1 and Time 3. MBSR training will be provided via an online website and secure data collection site called MySweetMind.org.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between the ages of 12 - 19
* Diagnosis of Type 1 Diabetes
* Fluent in English
* No diagnosed cognitive impairments
* 6th grade education completion
* Access to a Computer
* Access to the internet

Exclusion Criteria: under 12, over 19 - no access to a computer/internet

-

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2015-10-14 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-01-05 (Actual)

PRIMARY OUTCOMES:
Change in Mindful Attention Awareness Measurements after Mindfulness Training | Time 1 (Baseline), Time 2 (6 weeks post intervention) and Time 3 (3 months post intervention)
  Mindful Attention Awareness Adolescents Questionnaire developed by Brown, et al. (2011) to assess mindfulness in adolescents. The rapid increase in mindfulness based interventions for children and adolescents led the developers to modify the MAAS to measure mindfulness in this age group. It consists of 14 items that measure the level of mindfulness measured on a six-point scale with 1 (almost always) to 6 (almost never). Higher scores are an indication of more mindfulness in which there is a receptive state of mind to the present. The MAAS-A has been found to correlate with psychological well-being and healthy self-regulation and does measure the effects of mindfulness training. Mindful Attention Awareness will be measured three times to determine if there is a change in scores from Time 1 to Time 2 to Time 3
Change in Diabetes Quality of Life: DQOL-Y Measurements after Mindfulness Training | Time 1 (Baseline), Time 2 (6 weeks post intervention) and Time 3 (3 months post intervention)
  Diabetes Quality of Life - Youth Questionnaire (Ingersoll & Marrero, 1991) developed a modified version of the DQOL called the Diabetes Quality of Life for Youth (DQOL-Y). This questionnaire consists of 52 items with three subscales: Diabetes Life Satisfaction scale (17 items) with scores from 1 (very satisfied) to 5 (very dissatisfied), Disease Impact scale (23 items) with scores from 1 (never) to 5 (all the time), and Disease-Related Worries scale (11 items) with scores from 0 (does not apply) to 5 (all the time). Lower scores are indicative of higher quality of life. Also, included at the end is a general self-rating of overall health. In this study, quality of life was analyzed using the summation of each of these sub categories (impact, worry, and satisfaction to obtain a total DQOL score. Reliability of the DQOL-Y was tested for both adolescents and adults. The Diabetes Quality of Life questionnaire will be administered three times to determine whether or not there is a change
Change in HbA1c Measurements after Mindfulness Training | Time 1 (Baseline) and Time 3 (3 months post intervention)
  HbA1c measurement with fingerstick droplet of blood tested. The instant HbA1c required a drop of blood from the finger stick that provided results in less than 10 minutes. Less affected by the day to day variations in blood glucose readings, the HbA1c returns values which are representative of an average blood glucose over a 90 day period. The HbA1c will be administered two times to determine whether or not there is a change between Time 1 and Time 3.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Goodfellow, Study Chair — Duquesne University; Fran Cogen, MD, Study Director — George Washington University School of Medicine and Health Sciences; Jessica Devido, PhD, Study Director — Duquesne University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown KW, West AM, Loverich TM, Biegel GM. Assessing adolescent mindfulness: validation of an adapted Mindful Attention Awareness Scale in adolescent normative and psychiatric populations. Psychol Assess. 2011 Dec;23(4):1023-33. doi: 10.1037/a0021338. Epub 2011 Feb 14. PMID 21319908
- [Background] Ingersoll GM, Marrero DG. A modified quality-of-life measure for youths: psychometric properties. Diabetes Educ. 1991 Mar-Apr;17(2):114-8. doi: 10.1177/014572179101700219. PMID 1995281

DOCUMENTS (3):
  • Informed Consent Form: Parental Consent Form (2016-11-19): https://cdn.clinicaltrials.gov/large-docs/71/NCT03942471/ICF_000.pdf
  • Informed Consent Form: Consent Form Amended (2015-11-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT03942471/ICF_001.pdf
  • Study Protocol (2015-11-19): https://cdn.clinicaltrials.gov/large-docs/71/NCT03942471/Prot_002.pdf